CLINICAL TRIAL: NCT04230876
Title: Auditory Brain Training to Enhance Satisfaction and Usage of New Hearing Aids by Older Adults
Brief Title: Auditory Training and Hearing Aid Satisfaction
Acronym: ATandHAs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201909043
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Hearing Impairment, Sensorineural
Keywords: Auditory Training
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All participants experience the same interventions and assessments. Subjects are divided into either early or late intervention groups.
Who Masked: Participant
Masking Description: Participants are unaware if they are in the late or early intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Auditory Brian Training Games/Activities — Game-based activities that encourage listening to words and sentences in noisy situations. Participants will receive subscriptions to the clEAR online auditory training activities and recommended protocol for those who recently received new hearing aids.

SUMMARY:
Although hearing aids are the most common treatment for hearing loss, and have the potential to help seniors stay active and productive, almost 50% of them who receive hearing aids rarely if ever use them, a state of affairs sometimes referred to as "the hearing aid in the drawer" syndrome. clEAR's customized auditory brain training has been shown to be effective in improving adults' abilities to recognize speech, in reducing their perceptual effort associated with listening with a hearing loss, and in increasing their confidence to engage in everyday conversations. In the proposed research, we will determine whether older adults who receive hearing aids for the first time report higher satisfaction with their new hearing aids and have longer daily use time as a result of having completed clEAR's auditory brain training program for new hearing aid users.

DETAILED DESCRIPTION:
Auditory training as the potential to dramatically affect older persons' adjustment to a new hearing aid and to maximize the benefits they receive from wearing one. In turn, by wearing hearing aids, they experience easier and more successful communication patterns. They enhance their ability to engage in everyday conversations and will be able to become more socially involved with their family and friends. In this study we will try to determine the extent to which web-based clEAR auditory brain training, with concomitant support from a clEAR in-house audiologist, affects satisfaction with new hearing aids and increases daily use time. The study will include thirty adults over the age of 60 years who have received hearing aids for the first time. After an adjustment period, half will complete clEAR's auditory brain training program right away and the other half will complete it after a delay period, and both will complete a control condition. To establish the level of feasibility and clinical utility. We will measure hearing aid satisfaction, benefit ratings, and hearing aid use time.

ELIGIBILITY:
Inclusion Criteria:

* Must be a native English speaker
* Must have a mild to severe bilateral sensorineural hearing loss
* Must be a candidate for new hearing aid(s) (have never used hearing aids)

Exclusion Criteria:

* Cognitive impairment or any factors that would prohibit a participant from completing questionnaires
* Cognitive or speech production factors that would prohibit a participant from repeating words during a speech perception test.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The data collected are to be used exclusively by research team and clEAR.

RESULTS

PARTICIPANT FLOW:
Groups:
- Amptify First: The Amptify First group received the following order:
  1. Hearing aid adjustment period (2 weeks)
  2. The Amptify DTx curriculum, auditory training, and live coaching (4 weeks)
  3. Watch closed caption TV for 20 minutes each day (4 weeks)
- Amptify Second: The Amptify First group received the following order:
  1. Hearing aid adjustment period (2 weeks)
  2. Watch closed caption TV for 20 minutes each day (4 weeks)
  3. The Amptify DTx curriculum, auditory training, and live coaching (4 weeks)
Period: Overall Study
Arm/Group | Amptify First | Amptify Second
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — participant did not complete protocol by not training or not wearing aids. | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amptify First | Amptify Second | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.8 (7.0) | 70.3 (5.5) | 72.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Pure-Tone-Average [Mean (Standard Deviation); unit: Sound Level in dB(HL)]
  Right Ear | 30.4 (12.0) | 31.7 (11.7) | 31.4 (9.8)
  Left Ear | 32.5 (7.3) | 35.2 (9.1) | 33.5 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hearing Aid Satisfaction After Auditory Training
Description: The Client Orientated Scale of Improvement (COSI), a subjective measure of improvement on self-defined goals. The scale is relative to a baseline assessed before wearing hearing aids. For each goal participants select from a scale of improvement including Worse (-1), No Difference (0), Slightly Better (+1), Better (+2), and Much Better (+3). Positive values between one and three indicate improvement, negative values indicate that the self-defined goals got worse, and zero is no improvement. COSI scores were assessed before and after participants used the Amptify DTx. The outcome measure reported is the difference between scores before and scores after using the Amptify DTx.
Time Frame: Three weeks after hearing aid fitting and after completing the four week training protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amptify First | Amptify Second
Number analyzed (Participants) | 14 | 14
units on a scale | 1.9 (0.7) | 1.7 (0.9)
Statistical Analysis 1: Comparison: Amptify First vs Amptify Second; Test type: Superiority; p = 0.269, ANOVA — Within the 28 participants, changes in the COSI scores after four weeks using the Amptify were compared to the changes after four weeks watching 20 minutes of CC TV (F(1,26)=1.28); partial eta squared = 0.047

2. Primary Outcome: Change in Hearing Aid Satisfaction After Auditory Training
Description: The International Outcome Inventory for Hearing Aids (IOI-HA) is a hearing aid satisfaction questionnaire that averages a series of seven questions on a five-point scale (0-5 possible points of improvement). IOI-HA scores were assessed before and after participants used the Amptify DTx. The outcome measure reported is the difference between scores before and scores after using the Amptify DTx. Higher values between 1 and 5 indicate more relative satisfaction.
Time Frame: Three weeks after hearing aid fitting and after completing the four week training protocol.
Population: Two participants in the Amptify First group and one participant in the Amptify second group did not complete the first IOI-HA questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amptify First | Amptify Second
Number analyzed (Participants) | 12 | 13
units on a scale | 1.1 (0.4) | 0.1 (0.3)
Statistical Analysis 1: Comparison: Amptify First vs Amptify Second; Test type: Superiority; p = 0.401, ANOVA — Changes in the IOI-HA scores measured after four weeks using the Amptify were compared to the changes seen after four weeks of CC TV every day (F(1,23)=.733); partial eta squared = 0.031

3. Primary Outcome: Change in Hearing Aid Satisfaction After Auditory Training
Description: Abbreviated Profile of Hearing Aid Benefit (APHAB) is common clinical questionnaire for determining hearing aid benefit using a series of 24 questions on a seven-point scale (A-G; the scale is then converted to "percent of time" from 1% (Never) to 99% (Always) and 50% means half of the time). Hearing aid benefit is calculated as the difference between the performance with a hearing and and performance without a hearing aid. More positive values indicate more benefit.
Time Frame: Three weeks after hearing aid fitting and after completing the four week training protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amptify First | Amptify Second
Number analyzed (Participants) | 14 | 13
score on a scale | 17.4 (13.4) | 19.4 (12.3)
Statistical Analysis 1: Comparison: Amptify First vs Amptify Second; Test type: Superiority; p = 0.968, ANOVA — Changes in the APHAB benefit scores after four weeks using the Amptify were compared to the improvements seen after four weeks of CC TV every day (F(1,25)=.002); partial eta squared = 0.000

4. Primary Outcome: Change in Hearing Aid Satisfaction After Auditory Training
Description: The Speech, Spatial and Qualities of Hearing Scale (SSQ-12) is a subjective tool or assessing the quality of the sound from a hearing aid using a 12-item questionnaire. Questions focus on how well the participant could hear in various situations. The responses range on a scale from "Not At All" (0) to Perfectly (10). Higher values indicate better sound quality.
Time Frame: Three weeks after hearing aid fitting and after completing the four week training protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amptify First | Amptify Second
Number analyzed (Participants) | 14 | 14
units on a scale | 0.7 (2.7) | 0.5 (2.1)
Statistical Analysis 1: Comparison: Amptify First vs Amptify Second; Test type: Superiority; p = 0.392, ANOVA — Changes in the SSQ-12 scores after four weeks using the Amptify were compared to the improvements seen after four weeks watching 20 minutes of CC TV (F(1,26)=.756); partial eta squared = 0.028

5. Primary Outcome: Change in Hearing Aid Satisfaction After Auditory Training
Description: Daily use (in hours/day) is logged by the participant. Improvement is indicated by an increase in the amount of time the participant uses the hearing aid each day.
Time Frame: Three weeks after hearing aid fitting and after completing the four week training protocol.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Amptify First | Amptify Second
Number analyzed (Participants) | 14 | 14
hours/day | -.09 (2.3) | 0.8 (1.2)
Statistical Analysis 1: Comparison: Amptify First vs Amptify Second; Test type: Superiority; p = 0.720, ANOVA — Among the 28 participants, changes in the hours per day of hearing aid usage seen after four weeks using the Amptify were compared to the changes seen after four weeks of CC TV every day (F(1,26)=.131); partial eta squared = 0.005

6. Secondary Outcome: Change in Percent Words Correct on Speech Perception Measures After Auditory Training
Description: The NU-6 is a standard clinical assessment of word discrimination. Lists consist of 50 words in quiet and were presented through the Amptify DTx while wearing the hearing aid. NU-6 scores are in percent words correctly identified. Scores reported here are the difference between scores measured before and after completing the Amptify DTx.
Time Frame: At the time of hearing aid fitting (baseline), three weeks after hearing aid fitting, and after completing the four week training protocol.
Measure: Mean (Standard Deviation); unit: Percent words correct
Arm/Group | Amptify First | Amptify Second
Number analyzed (Participants) | 14 | 14
Percent words correct | 4.3 (7.8) | -1.0 (11.6)
Statistical Analysis 1: Comparison: Amptify First vs Amptify Second; Test type: Superiority; p = 0.242, ANOVA — Changes in the NU-6 seen after four weeks using the Amptify were compared to the changes seen after four weeks watching 20 minutes of CC TV (F(1,26)=1.43); partial eta squared = 0.052

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Amptify First | Amptify Second
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT04230876/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04230876/SAP_001.pdf
  • Informed Consent Form (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT04230876/ICF_002.pdf